CLINICAL TRIAL: NCT04926753
Title: Induction Chemotherapy Combined With Toripalimab in Locoregionally-Advanced Laryngo-Hypopharyngeal Squamous Cell Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhang, Chair of Department of Oncology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DETECTOR-1
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Locoregionally Advanced Laryngo-hypopharyngeal Squamous Cell Cancer
MeSH Terms: interventions — Fluorouracil; Cisplatin; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): 5-Fluorouracil(750 mg/m2/d, CIV d1-5) Cisplatin(75mg/m2,d1)/Carboplatin(AUC5, d1) Toripalimab 240mg d1
  Interventions: Drug: 5-Fluorouracil, Cisplatin, Toripalimab

INTERVENTIONS:
Drug: 5-Fluorouracil, Cisplatin, Toripalimab — Drug: FP combined with Toripalimab Combination drugs: 5-Fluorouracil(F), Cisplatin/Carboplatin(P) and Toripalimab every 21 days for 2 cycles This is a single-arm study with all patients receiving these three drugs.

SUMMARY:
This is a non-randomized phase 1, open-labeled clinical study, 1-arm, single center, to observe efficacy and safety of chemotherapy plus PD-L1 antibody Toripalimab every 21 days for 2 cycles as induction regimen in locoregionally-advanced laryngo-hypopharyngeal squamous cell cancer patients.

DETAILED DESCRIPTION:
Locoregionally advanced laryngo-hypopharyngeal squamous cell cancer patients have the demand of laryngo-preservation. Induction chemotherapy (FP) combined with Toripalimab (a humanized IgG4 monoclonal antibody against PD-1) will be given. This regimen will be given every 21 days for 2 cycles. Radiological examinations and PET(FDG/FAPI) examinations pre/post-treatment will be administrated for response evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients aged≥18 years.
2. Histologically confirmed Laryngo-hypopharyngeal squamous cell cancer, previously untreated (including surgery/radiotherapy/chemotherapy/immunotherapy).
3. Locoregionally-advanced disease stage cT2-4N0-3M0.
4. ECOG performance status 0 to 1.
5. Adequate organ function: Absolute neutrophil count (ANC) ≥1.5x109/L, White blood count ≥3.5x109/L, Platelets ≥75x109/L, Hemoglobin (Hb) ≥70g/L, ALT/AST ≤2.5x ULN (for patient with liver metastasis ALT/AST ≤5x ULN), Serum bilirubin ≤1.5x ULN, Serum creatinine ≤1.5x ULN.
6. HBV infected patients (inactive/asymptomatic carrier, chronic or active) with HBV DNA<500IU/ml (or 2500 copies/ml).
7. Pregnancy test of female patients with fertile activity should be negative within 7 days before enrollment. Patients should keep contraception during treatment.
8. Willingness and ability to comply with the protocol for the duration of the study including scheduled visits, examinations, investigations and treatment plans with informed consent form.

Exclusion Criteria:

1. Pregnancy or children bearing potential.
2. Metastasis.
3. Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
4. Have other malignant tumors within 5 years, except for fully treated basal cell/squamous cell skin cancer/cervical cancer
5. Uncontrolled clinical symptoms or diseases of the heart, such as: heart failure above NYHA II, unstable angina, myocardial infarction within 6 months;
6. With uncontrolled auto-immune diseases, interstitial pneumonia, ulcerative colitis, or patients who should receive long-term glucocorticoid treatment (>10mg/d prednisone).
7. With uncontrollable complications
8. Inadequate organ function
9. known hypersensitivity reaction to any of the study drugs or components.
10. Other unsuitable conditions determined by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 36 months

SECONDARY OUTCOMES:
Duration of response | 36 months
Progression free survival rate at 12 months | 12 months
Laryngo-preservation rate at 12 months | 12 months
Overall survival rate at 24 months | 24 months
Safety: adverse events as assessed by CTCAE v5. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Mingliang Xiang, MD & Ph.D, Principal Investigator — Ruijin Hospital; Jun Zhang, MD & Ph.D, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Oncology, Ruijin Hospital, Shanghai, China